CLINICAL TRIAL: NCT07041151
Title: Self-discontinuation of Urinary Catheters in Patients With Urinary Retention Following Gynecologic Surgery in a Rural Population
Brief Title: Self-discontinuation of Urinary Catheters in a Rural Population
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Ekaterina.A.Grebenyuk, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY02002854
Record Dates: First submitted 2025-06-18; First posted 2025-06-27 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Post-Operative Urinary Retention
Keywords: Post-operative urinary retention; Self-removal of foley catheter; Self-discontinuation of foley catheter; Post-operative void trial; Urogynecology; Pelvic surgery; Catheter management

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to either at-home foley catheter removal with a passive void trial or in-office catheter removal with a backfill void trial. Each participant will receive one intervention only and will be followed through postoperative recovery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- At-home passive void trial (Experimental): Participants will be instructed to remove their foley catheter at home 48-72 hours postoperatively. After removal, they will perform a passive void trial and will be monitored for successful voiding within a designated time frame. Instructions will be provided, and participants will be advised to contact the clinic if unable to void.
  Interventions: Other: At-home Foley Catheter Self-Removal with Passive Void Trial
- In-office backfill void trial (Active Comparator): Participants will return to the clinic 48-72 hours postoperatively for standard foley catheter removal and a backfill void trial. The bladder will be filled with 300 mL of sterile water, and voiding will be assessed in clinic per institutional protocol.
  Interventions: Other: In-Office Foley Catheter Removal and Backfill Void Trial

INTERVENTIONS:
Other: At-home Foley Catheter Self-Removal with Passive Void Trial — Participants will remove their foley catheter at home and perform a passive void trial. They will be instructed to drink fluids and attempt to void within a designated time frame. Instructions and support will be provided to ensure safety and follow-up, including clinic contact if voiding is unsuccessful.
  Arms: At-home passive void trial
Other: In-Office Foley Catheter Removal and Backfill Void Trial — Participants will return to clinic for removal of their foley catheter and undergo a backfill void trial. Standard protocols for instillation and assessment of urinary retention will be followed.
  Arms: In-office backfill void trial

SUMMARY:
The goal of this study is to understand patient satisfaction with two different ways of managing difficulty urinating after gynecologic surgery with a focus on those patients who receive care in a rural area.

One common practice is to have an "office catheter removal." This means, if a patient has trouble urinating after surgery and goes home with a foley catheter, they usually have to come back to the clinic within 2-3 days to have the catheter removed and to do a test to see if they can urinate on their own. For some patients, coming back to the clinic so soon after surgery can be difficult, especially for those patients who live far away or are dependent on others for getting to appointments.

A second, less common, practice is to have patients remove their own catheter at home, or "self-removal of urinary (Foley) catheter." With self-removal, patients remove their Foley catheter at home, and confirm that they are urinating normally. This approach has been shown to be safe, with similar patient satisfactions, and success, but those studies did not take into account situations where patients may live a rural area and/or travel a long distance to the medical center to receive care.

This study is comparing the in-office removal with self-removal. The goal is to find out which option patients prefer, how convenient each approach is, and how well they work. The main goal of this study is to understand patient satisfaction and improve care after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older
2. Undergoing gynecologic surgery with planned postoperative trial of void to confirm normal voiding prior to discharge home
3. Willing and able to provide informed consent
4. English-speaking
5. Willing to comply with study procedures, including follow-up phone calls and surveys

Exclusion Criteria:

1. Known urinary tract abnormalities (e.g., urethral strictures, neurogenic bladder) that may affect voiding.
2. Diagnosis of voiding dysfunction prior to surgery with need to self-catheterize.
3. Perioperative complication that necessitates indwelling catheter for a specific duration of time.
4. Joint surgeries that would affect ability to comply with study methods (e.g. that necessitates longer inpatient admission or reduces mobility beyond that normal for postop patients after gynecologic surgery)
5. Presence of significant cognitive or physical impairments that limit the ability to comply with study procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction with Void Trial Process | 2 weeks postoperatively
  Measured using a 0-100 mm visual analog scale (VAS) administered at the 2-week follow-up visit.

SECONDARY OUTCOMES:
Postoperative Urinary Retention | within 72 hours postoperatively
  Defined as inability to void ≥200 mL within 30 minutes after backfill (in-office) or failure to void minimum volume within 6 hours post-catheter removal (at-home).
Urinary tract infection | Within 30 days postoperatively
  Defined by positive urine culture (≥100,000 CFU/mL of uropathogen) and/or clinical diagnosis documented in the chart.
Adverse Events Related to Foley Catheter Removal or Void Trial | up to 30 days postoperatively
  Includes catheter reinsertion, pain, bleeding, ED visits, unplanned clinic visits, or other provider-documented complications.
Healthcare Resource Utilization | up to 30 days postoperatively
  Includes the number of MyDH messages, telephone encounters, and unplanned clinic or emergency department visits related to the void trial process, as documented in the electronic medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterina Grebenyuk, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (2):
- United States (2):
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Dartmouth Manchester Ambulatory Surgery Center, Manchester, New Hampshire

IPD SHARING:
Plan to Share IPD: No
This is a single-center, investigator-initiated study. There are no plans to share individual participant data at this time.